CLINICAL TRIAL: NCT05013905
Title: A Phase 2a, Multi-Center, Open-Label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of PRA023 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: A Phase 2a Safety and Efficacy Open-Label Study of PRA023 in Subjects With Moderately to Severely Active Crohn's Disease
Acronym: APOLLO-CD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prometheus Biosciences, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR200-103; 7240-006 (Other: MSD); 2023-509742-35-00 (Registry Identifier: EU CT); U1111-1309-6108 (Registry Identifier: UTN); 2021-000092-37 (EudraCT Number)
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
Keywords: APOLLO-CD; APOLLO; Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PRA023 (Experimental): Participants to receive PRA023 administered by intravenous (IV) infusion.
  Interventions: Drug: PRA023 IV; Device: Companion diagnostic (CDx)

INTERVENTIONS:
Drug: PRA023 IV — PRA023 administered at timepoints as directed by the protocol
  Other Names: PRA023 administered by IV Infusion
Device: Companion diagnostic (CDx) — CDx+ or CDx-

SUMMARY:
The purpose of this study is to assess the safety and efficacy of PRA023 in participants with moderately to severely active Crohn's Disease.

After the completion of the 12-week induction period, all participants have the option to continue in the open-label extension for another 38 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease
* Moderately to severely active CD as defined by Crohn's disease activity index (CDAI) score and centrally read endoscopy
* Must have corticosteroid dependence or have had no response, insufficient response, loss of response and/or intolerance to at least one of the following therapies: corticosteroid, immunosuppressants, or an approved anti-tumor necrosis factor (TNF), anti-integrin, or anti-interleukin (IL)12/23
* Able to provide written informed consent and understand and comply with the requirements of the study

Exclusion Criteria:

* Women of child bearing potential (WOCBP) and men with female partner of childbearing potential who are unwilling to use two highly effective methods of contraception to avoid pregnancy for the entire study period and up to 12 weeks after the last dose of study drug
* Diagnosis of ulcerative colitis (UC) or indeterminate colitis
* CD isolated to the stomach, duodenum, jejunum, or perianal region, without colonic and/or illeal involvement
* Suspected or diagnosed intra-abdominal or perianal abscess at screening
* Current stoma or need for colostomy or ileostomy
* Previous small bowel resection with a combined resected length of >100 cm or previous colonic resection of > 2 segments
* Surgical bowel resection within 3 months before screening
* Past or current evidence of definite low-grade or high-grade colonic dysplasia not completely removed
* Subjects in the opinion of the investigator are at an unacceptable risk for participation in the study
* Subjects who meet the protocol criteria for important laboratory exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2025-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prometheus Biosciences, Study Director — Clinicaltrials Call Center
Locations (34):
- United States (14):
  - Prometheus Biosciences Selected Site, Los Angeles, California
  - Prometheus Biosciences Selected Site, Liberty, Kansas
  - Prometheus Biosciences Selected Site, Chesterfield, Michigan
  - Prometheus Biosciences Selected Site, Ypsilanti, Michigan
  - Prometheus Biosciences Selected Site, St Louis, Missouri
  - Prometheus Biosciences Selected Site, Lebanon, New Hampshire
  - Prometheus Biosciences Selected Site, New York, New York
  - Prometheus Biosciences Selected Site, Garland, Texas
  - Prometheus Biosciences Selected Site, Lubbock, Texas
  - Prometheus Biosciences Selected Site, San Antonio, Texas
  - Prometheus Biosciences Selected Site, Southlake, Texas
  - Prometheus Biosciences Selected Site, Tyler, Texas
  - Prometheus Biosciences Selected Site, Bellevue, Washington
  - Prometheus Biosciences Selected Site, Tacoma, Washington
- Australia (3):
  - Prometheus Biosciences Selected Site, Bankstown, New South Wales
  - Prometheus Biosciences Selected Site, Woolloongabba, Queensland
  - Prometheus Biosciences Selected Site, Adelaide, South Australia
- Belgium (2):
  - Prometheus Biosciences Selected Site, Leuven
  - Prometheus Biosciences Selected Site, Liège
- Prometheus Biosciences Selected Site, London, Ontario, Canada
- Czechia (2):
  - Prometheus Biosciences Selected Site, Brno
  - Prometheus Biosciences Selected Site, Slaný
- France (4):
  - Prometheus Biosciences Selected Site, Clichy
  - Prometheus Biosciences Selected Site, Nice
  - Prometheus Biosciences Selected Site, Saint-Priest-en-Jarez
  - Prometheus Biosciences Selected Site, Vandœuvre-lès-Nancy
- Prometheus Biosciences Selected Site, Tbilisi, Georgia
- Poland (7):
  - Prometheus Biosciences Selected Center, Krakow
  - Prometheus Biosciences Selected Site, Rzeszów
  - Prometheus Biosciences Selected Site, Sopot
  - Prometheus Biosciences Selected Site, Torun
  - Prometheus Biosciences Selected Center, Warsaw
  - Prometheus Biosciences Selected Site, Warsaw
  - Prometheus Biosciences Selected Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Feagan BG, Sands BE, Siegel CA, Dubinsky MC, Longman RS, Sabino J, Laurent O, Luo A, Lu J, Nguyen DD, Munoz-Elias EJ, Llewellyn H, Wang Y, Jang I, Bilsborough J, Marchelletta R, Towfic F, Yen M, Anderson JK, DuVall A, Kierkus J, Woynarowski M, Al Kharrat H, Targan SR, McGovern DPB. Safety and efficacy of the anti-TL1A monoclonal antibody tulisokibart for Crohn's disease: a phase 2a induction trial. Lancet Gastroenterol Hepatol. 2025 Aug;10(8):715-725. doi: 10.1016/S2468-1253(25)00071-8. Epub 2025 May 30. PMID 40456235
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26174&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- PRA023: Participants received PRA023 administered by intravenous (IV) infusion as directed by the protocol.
Period: Overall Study
Arm/Group | PRA023
Started | 55
Completed | 53 (Completed Induction Period)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | PRA023
Number analyzed (Participants) | 55
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 18-44 years | 37
  Age (years): 45-64 years | 13
  Age (years): 65+ years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 48
  More than one race | 0
  Unknown or Not Reported | 4
Weight [Mean (Standard Deviation); unit: kg] | 77.6 (20.6)
Duration of Disease (years) [Mean (Standard Deviation); unit: years] | 10.29 (9.27)
Baseline Crohn's disease activity index (CDAI) Score [Mean (Standard Deviation); unit: score] — CDAI includes abdominal pain, stool frequency, general well-being, presence of complications (arthritis/arthralgia, uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI score is the sum of the 8 weighted scores and approximately ranges from 0 to 600; higher scores indicate more severe disease.
  score | 317.9 (67.2)
Number of Prior Exposure to Biologic Therapy [Count of Participants; unit: Participants]
  Biologic Naive | 16
  1 Prior Biologic | 10
  2 Prior Biologics | 10
  >=3 Prior Biologics | 19
Baseline Simple Endoscopic Score for Crohn's Disease (SES-CD) [Mean (Standard Deviation); unit: score] — Assessment of change in Simple Endoscopy Score for Crohn's Disease (SES-CD) from Baseline. Measure Description: The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
  score | 13.4 (6.7)
Concomitant Immunomodulator Use [Count of Participants; unit: Participants] | 8
Concomitant Oral Corticosteroid Use [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of participants who experienced treatment-emergent adverse events (AEs)
Time Frame: Week 12
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 43

2. Primary Outcome: Serious Adverse Events
Description: Number of participants who experienced serious adverse events (SAEs)
Time Frame: Week 12
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 8

3. Primary Outcome: Adverse Events Leading to Discontinuation
Description: Number of participants who experienced AEs leading to discontinuation
Time Frame: Week 12
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 2

4. Primary Outcome: Endoscopic Improvement
Description: Number of participants achieving induction of endoscopic improvement (decrease in simple endoscopy score for Crohn's disease [SES-CD] ≥ 50% from Baseline)
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores with no important protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 50
Participants | 13

5. Secondary Outcome: Clinical Remission
Description: Number of participants achieving clinical remission, as defined by Crohn's disease activity index [CDAI] score < 150
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 27

6. Secondary Outcome: Endoscopic and Clinical Improvement
Description: Number of participants who achieved a decrease in SES-CD ≥ 50% AND reduction in CDAI ≥ 100 points from Baseline or CDAI<150
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 9

7. Secondary Outcome: Number of Participants Achieving a Composite Response
Description: Composite response is defined as a decrease by at least 50% in hsCRP or fecal calprotectin from baseline and a reduction of either CDAI ≥ 100 points from Baseline or CDAI<150 in subjects with at least one elevated biomarker at baseline.
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores with at least one elevated biomarker at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 49
Participants | 17

8. Secondary Outcome: Normalization of C-reactive Protein
Description: Number of participants with normalization of hsCRP (as defined by hsCRP < 5 mg/L), among subjects with elevated concentrations at Baseline, at Week 12
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores who have elevated hsCRP values at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 36
Participants | 5

9. Secondary Outcome: Normalization of Fecal Calprotectin
Description: Number of participants with normalization of fecal calprotectin (fecal calprotectin < 250 ug/g), among subjects with elevated concentrations at Baseline, at Week 12
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores with elevated fecal calprotectin at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 44
Participants | 6

10. Secondary Outcome: Clinical Response
Description: Clinical response is defined as either a reduction of either CDAI ≥ 100 points from Baseline or CDAI<150.
Time Frame: Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 37

11. Secondary Outcome: Two Component Patient-reported Outcome (PRO-2) Remission
Description: Number of subjects with PRO-2 remission (defined as average daily abdominal pain score ≤ 1 point and average daily stool frequency ≤ 3 points with abdominal pain and stool frequency no worse than Baseline) at Week 12.
Time Frame: Week 12
Population: All subjects who have been treated with PRA023 with Baseline CDAI and SES-CD scores.
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 27

12. Secondary Outcome: Change From Baseline in Simple Endoscopy Score for Crohn's Disease (SES-CD)
Description: Assessment of change in simple endoscopy score for Crohn's Disease (SES-CD) from Baseline. Measure Description: The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy (ileum, right colon, transverse colon, sigmoid and left colon, and rectum). The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Baseline and Week 12
Population: All participants who have been treated with PRA023 with Baseline CDAI and SES-CD scores, who have SES-CD scores at Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRA023
Number analyzed (Participants) | 51
score on a scale | -2.6 (4.32)

13. Secondary Outcome: Serum Concentration of PRA023 (MK-7240)
Description: Blood samples were obtained for PK analysis of the serum concentration of PRA023 at week 12.
Time Frame: Week 12
Population: All participants who were treated with PRA023 with Baseline CDAI and SES-CD scores, and had blood samples drawn for serum concentration of PRA023
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PRA023
Number analyzed (Participants) | 53
ng/mL | 88199.1 (43811.21)

14. Secondary Outcome: Number of Participants Positive for Anti-drug Antibody (ADA)
Description: Blood samples were collected for the determination of anti-PR023 antibodies based on confirmatory assay. The number of participants with confirmed positive anti-PR023 antibodies results at any visit during the study is presented.
Time Frame: Up to approximately 12 weeks
Population: All participants who were treated with PRA023 with Baseline CDAI and SES-CD scores and had blood samples collected for ADA determination
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 55
Participants | 8

15. Secondary Outcome: Number of Participants With Positive Neutralizing Anti-Bodies (NAB)
Description: Blood samples were collected for the determination of NAB. The number of participants with positive NAB results at any visit during the study is presented.
Time Frame: Up to approximately 12 weeks
Population: All participants who were treated with PRA023 with Baseline CDAI and SES-CD scores and who were ADA positive post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PRA023
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Adverse event assessment occurred at every scheduled visit. An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Arm/Group | PRA023
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 8/55
Other Adverse Events (participants affected / at risk) | 20/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRA023 (N=55)
Crohn's Disease (Gastrointestinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 1
Anal Abscess (Infections and infestations) | 1
COVID-19 Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PRA023 (N=55)
COVID-19 (Infections and infestations) | 6
Urinary Tract Infection (Infections and infestations) | 5
Fatigue (General disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 4
Nasopharyngitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT05013905/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT05013905/SAP_001.pdf